CLINICAL TRIAL: NCT06261749
Title: Examination of Scapulothoracic Muscle Activation During Scapular Stabilizer Strengthening Exercises in the Prone Position with Voluntary Abdominal Contracture
Brief Title: Analysis of Scapular Musculature Activation During Targeted Abdominal Contraction with Scapular Stabilization Exercises
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Professor, Hacettepe University
Other Study IDs: EmgSCAPULA
Record Dates: First submitted 2024-01-19; First posted 2024-02-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-02

CONDITIONS: Scapula; Increased
Keywords: abdominal contractions; muscle activity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy individuals: Inclusion criteria:
  18-30 age Physical activity level should be at least 5 according to Tegner activity scale
  Interventions: Other: Voluntary Abdominal Contractions; Other: Exercise

INTERVENTIONS:
Other: Voluntary Abdominal Contractions — Abdominal contraction will be taught before exercise. They will be instructed to tighten their abdomen as if they were wearing tight pants and not to hold their breath. The visual biofeedback unit will be placed between the therapy table and the participant's abdominal area and will be used to monitor the contraction of the abdominal muscles. The visual biofeedback inelastic bag will be inflated to 70 mmHg and the participant will be instructed to draw the abdomen in and maintain the position. The participant will be asked to maintain a pressure of 60 mmHg during scapular retraction with visual feedback from an analog pressure gauge. Pressure changes of ± 5 mmHg due to breathing will be allowed. During exercise, the patient will be asked to perform the exercises while maintaining the pressure on the visual biofeedback.
Other: Exercise — Exercises;
  1. Scapular retraction with arms next to the trunk
  2. Scapular retraction with arms abducted at 45 degrees,
  3. Scapular retraction with arms 90 degrees abducted,
  4. Scapular retraction exercises with arms 120 degrees abducted The exercises will be performed with the shoulder head off the bed. The exercises will be repeated 3 times with 5 seconds rest between repetitions. To reduce the effect of fatigue, 2 minutes rest will be given between exercises. Each exercise will be performed with 3 seconds of concentric, 3 seconds of isometric and 3 seconds of eccentric contraction and muscle activation of UT-LT and SA muscles will be measured during these phases.

SUMMARY:
Muscle activation of the upper trapezius, lower trapezius and serratus anterior muscles will be measured during prone scapular retraction exercises. Then the same exercises will be performed with abdominal contraction using a stabilizer and muscle activity of the same muscles will be measured. A comparison will be made between the two conditions.

DETAILED DESCRIPTION:
The scapula plays an important role in providing both movement and stability of the shoulder joint. Correct scapular position and movement is achieved through the synchronized firing of muscles to provide optimal length-tension relationships between the scapular stabilizers. During arm elevation, coordinated muscle activation is seen between the serratus anterior (SA) and trapezius to provide controlled scapular upward rotation. Therefore, analyzing the muscle activation rates of these synergistic pairs (upper trapezius/serratus anterior [UT/SA] or upper trapezius/lower trapezius [UT/LT]) helps us understand scapular muscle function and prescribe exercises. Rehabilitation has focused on LT and SA muscle strengthening exercises to treat shoulder dysfunction . From a mechanical point of view, trunk and pelvis stability is required to transmit force and energy to the upper extremities during function or sports activities.

An altered spinal alignment directly affects the movement of the shoulder and scapular muscles, altering scapular position and stability. Coordinated activity of the shoulder and scapular muscles is essential to increase dynamic stability during shoulder movement; therefore, altered muscle activity can produce inappropriate glenohumeral and scapulothoracic joint movement rhythm and cause various shoulder pathologies examined the effect on the surface electromyographic activity of the scapulothoracic (UT, SA and LT) and middle deltoid muscles during isometric contraction in 45° shoulder abduction in the standing scapular plane supported by a pelvic and thoracic belt and reported that it did not significantly increase SA, LT activation, but increased middle deltoid activation and decreased UT electromyography activity observed an increase in the activity of the serratus anterior muscle during crossed shoulder flexion and scaption exercises with voluntary abdominal muscle contraction.

The resistance provided by isotonic exercise depends on gravity and the resistance pattern varies according to changes in the patient's body position (standing, prone, supine). In the prone position, it is often preferred because the scapular muscles can be strengthened in isolation by eliminating the lower extremity and core muscles. In a study in which trapezius muscle activation was examined by performing scapula retraction exercises in the prone position, a higher increase in trapezius muscle activation was reported compared to the standing study . It has been shown that there is a significantly greater increase in muscle activation in all 3 parts of the trapezius muscle in the prone position compared to the side lying and standing positions. It has been reported that this may be due to the fact that exercises performed prone against gravity may give more load to the trapezius muscle than the standing position. Although lower extremity movements are limited in the prone position compared to the standing position, anterior pelvic tilt formation as a result of excessive lumbar spine movements during exercises performed in this position should not be overlooked.

Therefore, our aim in this study was to investigate scapulothoracic muscle activations during open kinetic chain strengthening exercises with scapular stabilizers by providing lumbopelvic stability with voluntary abdominal contraction in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18-30
* Physical activity level of at least 5 on the Tegner activity scale.

Exclusion Criteria:

* Having pathology of the shoulder and spine
* History of previous upper extremity surgery
* Body mass index greater than 24.9
* Experience with core stability training.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include 30 healthy participants regardless of gender.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Electromyography | initial assesment (baseline)
  An 8-channel surface electromyography system will be used to measure muscle activation levels. A synchronized video recording will be taken.
  Electrode placement and inter-electrode distance will follow the recommendations of "Surface ElectroMyography for Non-Invasive Assesment of Muscles" (SENIAM), and bipolar silver/silver chloride surface electrodes will be placed with an inter-electrode distance of 2 cm. For UT, the electrodes will be placed between the C7 spinal vertebra and the posterior acromion; for AT, the electrodes will be placed at the 2/3 point of the line between the trigonum spinae and the T8 spinal vertebra; for SA, the electrodes will be placed horizontally just below the axillary region, at the level of the lower end of the scapula and medial to the latissimus dorsi.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Çaylan Gürses, Principal Investigator — Hacettepe University; İrem Düzgün, Study Director — Hacettepe University; Özgün Uysal, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided